CLINICAL TRIAL: NCT06370559
Title: The Relationship Between Repetitive Negative Thinking (RNT) and CBT Treatment Outcome Within a Specialist Anxiety Disorders Clinic.
Brief Title: Relationship Between Repetitive Negative Thinking and CBT Outcomes
Status: Completed | Type: Observational
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 339042
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anxiety Disorders; Obsessive-Compulsive Disorder; Post-traumatic Stress Disorder; Social Anxiety Disorder; Specific Phobia; Panic Disorder; Body Dysmorphic Disorders
Keywords: Rumination; Ruminative Thinking Questionnaire (RTQ-10); Cognitive Beavioural Therapy (CBT); Outcomes
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Phobia, Social; Phobia, Specific; Panic Disorder; Body Dysmorphic Disorders; Rumination Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the role of repetitive negative thinking (measured by the RTQ) in adult populations from an anxiety disorders and trauma clinic.

The main questions it aims to answer are:

* Whether the repetitive negative thinking can be used to predict i. initial symptom severity, and ii. therapy outcome (measured by change in scores on disorder specific measures).
* Whether change in RTQ mediates change in outcome Participants are sent weekly questionnaires that measure their progress. Within these questionnaires are the RTQ and other disorder-specific measures that we will be analysing.

Researchers may also compare clients with different disorders to see the accuracy the RTQ can predict treatment outcomes for each disorder.

DETAILED DESCRIPTION:
We are looking to examine how repetitive negative thinking (RNT; i.e. rumination and worry), measured by the repetitive thinking questionnaire (RTQ), affects the outcomes of Cognitive Behavioural Therapy (CBT) for anxiety and trauma disorders. Our study will involve looking over data collected from clients who completed treatment at the Centre for Anxiety Disorders and Trauma (CADAT) from 01/01/2022 to 31/03/2024, we will look at data from before they started treatment, whilst in treatment and once they completed treatment. This is an important issue to address as there is little guidance within existing CBT protocols on to how to identify and target RNT during treatment. Evidence also suggests that not only does RNT maintain anxiety disorders, but it can also interfere with therapy outcome. Research has found that patients receiving CBT for PTSD who displayed high-levels of rumination within their early CBT sessions had poorer outcomes in therapy. Our aim is to formally analyse the relationship between scores on the RTQ and both symptom severity and CBT treatment outcome for anxiety disorders. This would help us to test our hypotheses about the relationship (i.e. those with high RNT have poorer treatment outcomes and changes in RNT predict outcome across a range of anxiety and trauma disorders) and provide a basis for augmenting our existing treatments with interventions that specifically target this process.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed a course of CBT treatment at CADAT for one of the following anxiety disorders: OCD, PTSD, Panic Disorder, Health Anxiety, Emetophobia, Specific Phobia, Social Phobia, BDD, GAD, DPD or Hoarding.
* Participants must have completed regular questionnaires throughout their treatment.

Exclusion Criteria:

* Participants who dropped out of treatment
* Participants who did not complete online questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our sample consists of clients who have completed a course of CBT treatment from the Centre of Anxiety Disorders and Trauma between 01/01/2022 to 01/02/2024. Patients are typically seen for 12-20 sessions.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Repetitive Ruminative Thinking Questionnaire score | From pre treatment to post treatment for CBT at CADAT (an average of 12-20 weeks)
  Change in RTQ from pre- to post-treatment
Change in disorder-specific measure score | From pre treatment to post treatment for CBT at CADAT (an average of 12-20 weeks)
  Change in disorder-specific measure scores from pre- to post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Anxiety Disorders and Trauma, London, United Kingdom